CLINICAL TRIAL: NCT06504303
Title: Comparison of Socket Geometry and Clinical Outcomes Between Manually- and Digitally-designed Prosthetic Sockets for Lower-limb Amputees: a Feasibility Study
Brief Title: Socket Geometry and Clinical Outcomes of Manual vs Digital Sockets for Lower-limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-013-WP
Record Dates: First submitted 2021-07-28; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Amputation
Keywords: Transtibial amputation; Prosthesis; 3D printing; Additive manufacturing; Computer-aided design; Socket Comfort Score

STUDY DESIGN:
Intervention Model Description: Participants will be measured for a prosthetic device through (1) manual casting using Plaster of Paris bandages and (2) scanning using a 3D scanner. Subjects will be given a patient experience survey to score their experience with each shape capturing process. Two sockets, one made from each of the two shape-capturing methods, will be 3D printed.
  Both sockets will be fitted to the subject. The immediate socket fit will be recorded by the number of filler sock plys needed to be added in the socket. Subjects will continue therapy using the socket that is more comfortable and fits better, based on both the subject's judgment and the judgment of their clinician. If the subject finds both sockets as equally comfortable, he/she will get to choose the preferred socket to continue with for therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D-printed socket (Experimental): The 3D scan of the participant's residual limb will be digitally-modified and fabricated using 3D printing.
  Interventions: Device: 3D-printed socket

INTERVENTIONS:
Device: 3D-printed socket — During the shape-capturing in-patient appointment, participants will be measured for the prosthetic device through (1) manual casting using Plaster of Paris bandages and (2) scanning using a 3D scanner. The clinician will manually modify the positive plaster cast and digitally modify the scanned impression using OMEGA software. The manually-modified positive cast will be digitized by scanning the cast, then 3D-printed. The digitally-modified socket file will also be 3D printed. The research investigator will make a de-identified mark on each socket to differentiate between the two sockets after 3D printing, and will record the order in which the sockets are fit to the patient.

SUMMARY:
The most important aspect of a lower-limb prosthesis is the socket as the interface between the human and the mechanical prosthetic system. Proper fit of the socket to the residual limb is a critical factor in determining comfort, suspension, energy expenditure and ultimately the functional efficiency of the remaining prosthesis. Patients may not wear their prosthesis if they find the socket uncomfortable.

Traditional manufacturing of prosthetic sockets is a high-skill process involving several stages. Capturing the shape of the residual limb and modifying the mould is performed with a manual, hands-on approach. This leads to inconsistencies between clinicians, and increases the likelihood of human error. There is opportunity to improve this process with advanced computer-aided design (CAD) and manufacturing (CAM). 3D printing can be leveraged for its ability to effortlessly manufacture one-off, complex and organic shapes, such as prosthetic sockets. However, the digital method removes the tactile feedback that the clinician generally benefits from when manually designing the socket, thus leading to some uncertainty in how they are modifying the socket. Moreover, the difference in the learning curve may cause inconsistencies in modifications made by different clinicians.

While clinicians may be hesitant in their knowledge-transfer from a manual to digital method, sockets designed using CAD still produce successful outcomes. To facilitate wider-spread adoption of 3D printing as a standard tool in the clinic, more research is needed to better understand how the digital design process affects the geometry of the socket, and how this affects clinical outcomes for amputees.

The investigators hypothesize that (1) digitally-designed sockets and manually-designed sockets will have geometric differences, (2) the digitally-designed socket will result in better clinical outcomes compared to manually-designed sockets, and (3) improved clinical outcomes will correlate to geometric differences centred on particular regions of the socket. However, a feasibility study is needed to inform an effective protocol. This feasibility study aims to explore socket geometries and prosthetic outcomes compared between manually-designed and digitally-designed devices for lower-limb amputees. Findings will help in improving the current 3D printing techniques and exploring outcomes for the users.

DETAILED DESCRIPTION:
This crossover case-control feasibility study aims to explore socket geometries and prosthetic outcomes compared between manually-designed and digitally-designed devices for lower-limb amputees. Feasibility and outcome measures will be measured at three major stages of routine prosthetic care, namely the socket fabrication, socket fitting, and functional testing.

Socket Fabrication:

Participants will be measured for the prosthetic device through (1) manual casting using Plaster of Paris bandages and (2) scanning using a 3D scanner (Artec Eva, Artec 3D, Luxembourg). The patient's residual limb soft tissue density will also be measured using a standard gauge (Fowler depth gage, Fowler Co., Inc., Massachusetts, USA) on certain landmarks: medial flare, distal end, lateral, popliteal region, distal tibia. The clinician will manually modify the positive plaster cast (herein, the M-socket) and digitally modify the scanned impression (herein, the AD-socket) using OMEGA software (OMEGA software, WillowWood Global LLC, Ohio, USA). The M-socket positive cast will be digitized by scanning the cast and exporting it to OMEGA. This scanned M-socket file and the CAD-socket file will each be 3D printed (Stratasys F370, Stratasys Ltd., Minnesota, USA) in nylon-based thermoplastic. Conventionally, the socket is manufactured by draping thermoplastic over a mold, but for this study, both sockets will be 3D printed. The two 3D-printed sockets will then be reinforced and connected to its corresponding component adapters using fiberglass and resin materials, as is done during current standard of care. To eliminate confounding, the same suspension and components will be used. Subjects will be given a patient experience survey to score their experience with each shape capturing process. The survey will be administered by a research assistant using a face-to-face interview technique before they are fit with the sockets.

Socket Fitting:

Both sockets will be fitted to the subject and immediate Socket Comfort Score will be recorded through an analogue visual scale, and will be recorded for every day that the patient wears each device. The immediate socket fit will be recorded by the number of filler sock plys needed to be added in the socket. Also, changes made to the sockets by the clinician (e.g., spot relieving) will be recorded. Subjects will continue therapy using the socket that is more comfortable and fits better, based on both the subject's judgment and the judgment of their clinician. If the subject finds both sockets as equally comfortable, he/she will get to choose the preferred socket to continue with for therapy. A healthcare provider will assist in the selection, should the patient request it. The subjects will be given 2 days to acclimate to the selected socket and will be retested for Socket Comfort Score once a day during the subject's therapy sessions, and tested for function one day before discharge (defined below).

Functional Testing:

One day before discharge from West Park, upon the completion of therapy, the participants will be tested for function through the L-test and 2-minute walk test (2MWT). This timeline is to ensure that the participant is safe to walk outside the parallel bars. The L test of functional mobility will be administered with the device. For patient safety, chairs will be placed in close proximity to the testing area, and subjects are allowed to walk with a mobility aid of their choice. One practice run will be allowed, followed by 2 trials with a 1-minute rest between trials. The mean times from the 2 trials will be used for data analysis. As a second measure of function, a 2-minute walk test (2MWT) will be administered after the L-test. To control for learning and practice effects, the subjects will be familiar with the test, or given 1 or more practice tests at least 1 day before testing. Subjects are allowed to walk with a mobility aid of their choice and allowed to rest during the 2-minute time.

The functional tests will be performed in the order described. The functional data will be collected by a member of the team other than the clinician that fits the patient in order to prevent bias in the results. Tests will be administered by a physiotherapist who is not involved in the study to ensure patient safety. To blind the device, the investigators will not disclose to the patient about the method the socket was designed when they first trial it. After the completion of the study, the participant will take the device home.

Clinical outcome measure data will be reported descriptively (mean, SD, minimum and maximum), and a statistical analysis plan detailing intended analyses will be drafted before the completion of data collection to inform a future study. The effect size will be calculated to help support sample size calculations for a future study. Feasibility data will be collected, and success of the feasibility analysis will be determined based on the following a priori criteria: recruitment rate ≥70% of all eligible potential participants; of the participants recruited, ≥70% adhered to the described protocol allowing for effective collection of quantitative and qualitative data appropriate for use in a definitive study; <20% dropped out of the study; SCS, L-test and 2MWT were identified as acceptable and appropriate outcome measures for the protocol; quantitative and qualitative data implied that digitally-designed sockets have different geometries to manually-designed sockets. Recruitment, adherence and drop-out rates will be calculated using the average obtained between the start of the study (once active recruitment starts) and the end of the study (once the desired sample size is reached). This study will decide that a larger study is not feasible if at least one of the criteria is not met.

ELIGIBILITY:
Inclusion Criteria:

* In-patient adults (18 years and older)
* Unilateral transtibial amputation
* Eligible to receive a preparatory prosthetic device
* Able to communicate in English orally and in writing
* Able to tolerate participating in an additional 30- minute 3D scanning session

Exclusion Criteria:

* Presentation of significant cognitive impairment
* History of epilepsy
* On dialysis at any point of the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Patient recruitment rates | Through study completion, an average of 1 year
  The number of eligible vs. recruited patients will be tracked throughout the study period.
Adherence to protocol | Through study completion, an average of 1 year
  Adherence to protocol steps (i.e., casting, CAD, 3D printing, or functional testing protocols) will be tracked throughout the study period and a standardized checklist of procedures will be kept to measure the rate at which procedures are implemented as intended for fidelity assessment.
Patient retention rates | Through study completion, an average of 1 year
  Patient drop-out rate will be tracked throughout the study period.

SECONDARY OUTCOMES:
Socket geometric differences | Through study completion, an average of 1 year
  The 3D geometries of the two sockets will be compared by superimposing the two files in CAD software and measuring the dimensional variances over the entire impressions. Global average difference, and local differences at anatomical areas where rectifications are made will be recorded. These include pressure sensitive areas of the patella, tibial tuberosity, distal tibia, fibular head, and medial and lateral femoral condyle; and pressure tolerant areas of the patellar tendon, medial and lateral flare of tibia, lateral flare of fibula, popliteal area, and distal end of stump. Any other major differences that are identified will be measured and their location recorded.
Socket comfort score change | Through study completion, an average of 1 year
  A numeric scale to capture socket comfort by patients will also be used (0 = not at all comfortable; 10 = very comfortable).
Two-minute walk test | Performed one day prior to discharge from West Park.
  Participants will be instructed to walk back and forth, as far as they can in 2 minutes without any further encouragement. One or more practice tests are allowed at least one day before testing. The test administrator will walk behind the subject to minimize the effect of pacing.
L-test | Through study completion, an average of 1 year
  Participants will be instructed to stand up from the chair, walk straight forward 7 meters, turn 90 degrees, walk 3 meters, turn 180 degrees and return to sit in the chair. A stopwatch will be used to record the time from the word 'go' to when the subject's buttocks first hits the seat surface when they return. The test administrator will use a digital stopwatch to time and a calibrated wheel with a counter to measure the distance walked. One practice run is allowed, followed by 2 trials with a 1-minute rest between trials. The mean times from the 2 trials will be used for data analysis.

OTHER OUTCOMES:
Demographics | Through study completion, an average of 1 year
  Demographic questions collected from people with LLAs will include: age, sex, cause of amputation, level of education, and work status.
Physiological Cost Index | Through study completion, an average of 1 year
  Calculated from two-minute walk test heart rates as the difference between resting and active heart rates, divided by the average walking speed based on the distance walked over the 2 minutes. The PCI correlates well with oxygen uptake in amputees, and therefore provides a useful estimate of walking efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Heim, MSc, C.P.(c), Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No